CLINICAL TRIAL: NCT02520414
Title: A Pilot Study to Assess the Feasibility of the Symphion® Bipolar Hysteroscopic Tissue Resection System in an Office Environment
Brief Title: Symphion® System In-Office Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minerva Surgical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U0524
Record Dates: First submitted 2014-11-06; First posted 2015-08-11 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Uterine Leiomyomas; Endometrial Polyps
MeSH Terms: conditions — Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Symphion® (Experimental): Patients treated in-office with Symphion® Bipolar Hysteroscopic Tissue Resection System.
  Interventions: Device: Symphion® Bipolar Hysteroscopic Tissue Resection System

INTERVENTIONS:
Device: Symphion® Bipolar Hysteroscopic Tissue Resection System

SUMMARY:
The purpose of this study is to determine the safety and feasibility of using the Symphion system in an office setting.

DETAILED DESCRIPTION:
The purpose is to determine the safety and feasibility of using an intrauterine tissue resection system in the office setting, as well as to expand the national discussion regarding in-office hysteroscopic procedures as it relates to the highest standards of care and cost containment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the approved Instructions for Use for the Symphion® bipolar hysteroscopic tissue resection system
* Confirmation hysteroscopic evaluation to access appropriate pathology type and size meets the Protocol guidelines for inclusion
* Subject has signed written Informed Consent

Exclusion Criteria:

* Subjects who are pregnant
* Subjects who have an active genital tract infection (as assessed by the physician)
* Subjects who have cervical malignancies
* Subjects who have previously been diagnosed with endometrial cancer
* Subjects who have Type 2 intracavitary myomas
* Type 0 or 1 intracavitary myoma greater than 3.0 cm

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Women's Surgery, Albuquerque, New Mexico, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Symphion®: Patients treated in-office with Symphion® Bipolar Hysteroscopic Tissue Resection System.
  Symphion® Bipolar Hysteroscopic Tissue Resection System
Period: Overall Study
Arm/Group | Symphion®
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Symphion®
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (7.2)

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of the Symphion® Bipolar Hysteroscopic Tissue Resection System When Used in the Office Setting for the Removal of Intracavitary Polyps and Myomas.
Description: Absence of device related adverse events, or death.
Time Frame: 2 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Symphion®
Number analyzed (Participants) | 10
percentage of participants
  Adverse Events | 0
  Device Malfunctions | 0

ADVERSE EVENTS:
Arm/Group | Symphion®
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No